CLINICAL TRIAL: NCT06230224
Title: A Phase 3, Randomized, Open Label Study Evaluating the Efficacy and Safety of Odronextamab (REGN1979), an Anti-CD20 x Anti-CD3 Bispecific Antibody, Versus Standard of Care Therapy in Participants With Relapsed/Refractory Aggressive B-cell Non-Hodgkin Lymphoma (OLYMPIA-4)
Brief Title: A Trial to Learn How Effective and Safe Odronextamab is Compared to Standard of Care for Adult Participants With Previously Treated Aggressive B-cell Non-Hodgkin Lymphoma
Acronym: OLYMPIA-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-HM-2299; 2022-502783-21-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2023-12-29; First posted 2024-01-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: B-Cell Non-Hodgkin Lymphoma (B-NHL)
Keywords: Non-Hodgkin lymphomas (NHLs); Aggressive NHL; B-Cell Non-Hodgkin Lymphoma (B-NHL); Odronextamab; Anti-CD20 × anti-CD3 bispecific antibody; Relapsed/Refractory NHL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — Ifosfamide; Carboplatin; Etoposide; etoposide phosphate; Rituximab; Dexamethasone; Calcium Dobesilate; Cisplatin; Cytarabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Odronextamab (Experimental): Participants will receive odronextamab monotherapy.
  Interventions: Drug: Odronextamab
- Standard Of Care (Active Comparator): Participants will receive salvage therapy (ifosfamide, carboplatin, etoposide ± rituximab [ICE ± R], or dexamethasone, cisplatin, cytarabine ± rituximab [DHAP ± R], or gemcitabine, dexamethasone, cisplatin ± rituximab [GDP ± R]) and continue with autologous stem cell transplant (ASCT) following a complete response (CR)/partial response (PR).
  Interventions: Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Rituximab; Drug: Dexamethasone; Drug: Cisplatin; Drug: Cytarabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Odronextamab — Administered by intravenous (IV) infusion
  Other Names: R1979
  Arms: Odronextamab
Drug: Ifosfamide — Administered by IV infusion, as part of the ICE ± R salvage therapy
  Other Names: Ifex
  Arms: Standard Of Care
Drug: Carboplatin — Administered by IV infusion, as part of the ICE ± R salvage therapy
  Other Names: Paraplatin
  Arms: Standard Of Care
Drug: Etoposide — Administered by IV infusion, as part of the ICE ± R salvage therapy
  Other Names: Etopophos
  Arms: Standard Of Care
Drug: Rituximab — Administered by IV infusion, as part of the ICE ± R, or DHAP ± R, or GDP ± R salvage therapy.
  Other Names: Rituxan
  Arms: Standard Of Care
Drug: Dexamethasone — Administered by IV, or orally (PO) as part of the DHAP ± R, or GDP ± R salvage therapy.
  Other Names: Decadron
  Arms: Standard Of Care
Drug: Cisplatin — Administered by IV infusion, as part of the DHAP ± R or GDP +/-R salvage therapy.
  Other Names: Platinol
  Arms: Standard Of Care
Drug: Cytarabine — Administered by IV infusion, as part of the DHAP ± R salvage therapy.
  Other Names: Cytosar-U
  Arms: Standard Of Care
Drug: Gemcitabine — Administered by IV infusion, as part of the GDP ± R salvage therapy.
  Other Names: Gemzar
  Arms: Standard Of Care

SUMMARY:
This study is researching an experimental drug called odronextamab, referred to as study drug. The study is focused on patients with previously treated aggressive B-cell non-Hodgkin lymphoma whose cancer has stopped responding to treatment (also known as 'refractory') or has returned (also known as 'relapsed'). The aim of the study is to see how safe, tolerable and effective the study drug is when given alone.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug versus Standard of Care (SOC)
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)
* Comparing the impact from the study drug versus SOC on quality-of-life and ability to complete routine daily activities

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically proven aggressive B-NHL, as described in the protocol. Availability of tumor tissue for submission to central laboratory is required for study enrollment. Archival tumor tissue for histological assessment prior to enrollment is allowed
2. Have primary refractory or relapse 12 months or less (≤) from initiation of frontline therapy Only patients who received 1 prior line of therapy containing an anti-Cluster of Differentiation 20 (CD20) antibody and anthracycline are allowed for enrollment
3. Have measurable disease with at least one nodal lesion with longer diameter (LDi) greater than 1.5 cm or at least one extranodal lesion with LDi greater than 1.0 cm, documented by diagnostic imaging (computed tomography [CT] or magnetic resonance imaging [MRI])
4. Intent to proceed to autologous stem cell transplant (ASCT), as described in the protocol
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
6. Adequate hematologic and organ function.

Key Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known involvement by non-primary CNS NHL, as described in the protocol
2. History of or current relevant CNS pathology, as described in the protocol
3. A malignancy other than NHL unless the participant is adequately and definitively treated and is cancer free for at least 3 years, with the exception of localized prostate cancer, cervical carcinoma in situ, breast cancer in situ, or nonmelanoma skin cancer that was definitively treated
4. Any other significant active disease or medical condition that could interfere with the conduct of the study or put the participant at significant risk, as described in the protocol
5. Wash-out period from prior anti-lymphoma treatments and infections, as described in the protocol
6. Allergy/hypersensitivity to study drug, or excipients.

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-05-14 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) as assessed by independent central review (ICR) | Assessed up to 3 years

SECONDARY OUTCOMES:
Progression free survival (PFS) as assessed by ICR | Assessed up to 3 years
Best overall response (BOR) as assessed by ICR | Assessed up to 6 months
Overall survival (OS) | Assessed up to 3 years
Overall change in physical functioning as measured by scores of the physical function scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC-QLQ-C30) | Assessed up to 3 years
  The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
EFS as assessed by local investigator | Assessed up to 3 years
PFS as assessed by local investigator | Assessed up to 3 years
BOR as assessed by local investigator | Assessed up to 6 months
Complete response (CR) as assessed by ICR | Assessed up to 6 months
CR as assessed by local investigator | Assessed up to 6 months
Duration of response (DOR) assessed by ICR | Assessed up to 3 years
DOR assessed by local investigator | Assessed up to 3 years
Incidence of treatment-emergent adverse events (TEAEs) | Assessed up to 1 year
Severity of TEAEs | Assessed up to 1 year
Odronextamab concentrations in serum | Assessed up to 6 months
Incidence of anti-drug antibodies (ADAs) to odronextamab over the study duration | Assessed up to 6 months
Titers of ADAs to odronextamab over the study duration | Assessed up to 6 months
Incidence of neutralizing antibodies (NAb) to odronextamab over the study duration | Assessed up to 6 months
Measurable residual disease (MRD) status | Assessed up to 6 months
Overall change in patient-reported outcomes (PROs), as measured by scores of the EORTCQLQ- C30 | Assessed up to 3 years
  The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Overall change in PROs, as measured by scores of the Functional Assessment of Cancer Therapy-Lymphoma (FACT-LymS) | Assessed up to 3 years
  The FACT-Lym lymphoma subscale (LymS) includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Overall change in PROs, as measured by scores of the EuroQol-5 Dimension-5 Level Scale (EQ-5D-5L) | Assessed up to 3 years
  The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Overall change in score of the Global Population item 5 (GP5) of the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire | Assessed up to 3 years
  A single item GP5 of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (99):
- Argentina (8):
  - Hospital Aleman, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundaleu - Fundacion Para Combatir La Leucemia, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Hospital Privado Universitario de Cordoba, Córdoba
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Olivia Newton John Cancer Wellness & Research Centre, Heidelberg, Victoria
- Brazil (15):
  - Hospital Santa Izabel - Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Ensino e Terapia de Inovacao Clinica Amo (Etica), Salvador, Estado de Bahia
  - Hospital Sirio Libanes Brasilia, Brasília, Federal District
  - Uopeccan Hospital do Cancer de Cascavel, Cascavel, Paraná
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado, Porto Alegre, Rio Grande do Sul
  - Amaral Carvalho Hospital, Jaú, São Paulo
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
  - A Beneficencia Portuguesa de Sao Paulo, Oncology House, São Paulo
  - Instituto D'Or De Pesquisa e Ensino, São Paulo
  - Hospital das Clinicas, Faculty of Medicine, University of Sao Paulo, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
- Chile (2):
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan
- Colombia (2):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Clinica Imbanaco, Cali, Valle del Cauca Department
- Hungary (2):
  - University of Pecs, Pécs, Baranya
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-Cesena
  - Centro Di Riferimento Oncologico (CRO), Aviano, National Cancer Institute, Aviano, Pordenone
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - AOU Maggiore della Carita, Novara
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese
- Malaysia (5):
  - Hospital Sultanah Aminah Jhor Bahru, Johor Bahru, Johor
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Kuala Lumpur, Selangor
  - Subang Jaya Medical Center, Subang Jaya, Selangor
- Erasmus University Medical Center, Rotterdam, Netherlands
- Romania (2):
  - Coltea Clinical Hospital, Bucharest, București
  - Ion Chiricuta Oncology Institute, Cluj-Napoca, Cluj
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
- South Korea (13):
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - St. Vincent Hospital - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeyungnam University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Asan Medical Center, Seoul
  - Seoul St Marys Hospital, Seoul
  - Yeouido St. Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Virgen De Las Nieves De Granada, Granada
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Clinica Universidad de Navarra- Pamplona, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
  - University Hospital Doctor Peset, Valencia
- Taiwan (11):
  - Chang Gung Medical Foundation, Chiayi City, Chianan Plain
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District, Hunan Province
  - Changhua Christian Hospital, Changhua
  - Show Chwan Memorial Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Taichung General Veterans Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Chulalongkorn University, Bangkok
  - Sriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (11):
  - Ankara University Faculty of Medicine, Mamak, Ankara
  - Gazi University, Ankara, Central Anatolia
  - VM Medical Park Mersin Hospital, Mezitli, Mersin
  - Tekirdag Namik Kemal University Hospital, Tekirdağ, Suleymanpasa
  - Sbu Dr.A.Y. Ankara Onkoloji Suam, Ankara
  - VKV American Hopital, Istanbul
  - Istanbul University, Istanbul
  - Ege University, Izmir
  - Sakarya University Medical Faculty, Sakarya
  - Ondokuz Mayıs University, Samsun
  - Zonguldak Bulent Ecevit University, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: OLYMPIA — https://olympiastudies.com/en-us